CLINICAL TRIAL: NCT07341932
Title: Helium-free Magnetocardiography Guided Therapy for Stable Coronary Artery Disease - A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, song xiantao, Director of Cardiology Ward A, Department of Cardiology I, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024AZB1003; 2024AZB1003 (Other Grant/Funding Number: Beijing Anzhen Hosptial, Capital Medical University)
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Stable Coronary Artery Disease CAD
Keywords: Stable coronary artery disease CAD; MCG; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Allocation concealment was implemented using a web-based central randomization system. Study site staff entered each participant's basic information (initials, age, gender, subject ID, etc.) and stratification factors into the system. Based on the predefined principles, the system automatically generated a unique random number and subject ID, and notified the investigator at the respective site via the network regarding the participant's assignment to either the intervention or control group. Upon receiving the randomization result, the site investigator administered the corresponding treatment-either the intervention or control therapy-according to the assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Management Group (Experimental): Treatment strategies were recommended based on stenosis severity, pre-test probability, and functional test results: For patients with 50-70% stenosis, if the pre-test probability was <15%, treatment recommendations had to be made by clinicians integrating one or more functional test results (e.g., exercise ECG, stress echocardiography, SPECT, stress CMR); if the pre-test probability was ≥15%, it was advised to recommend treatment strategies considering functional test results. For patients with CCTA-indicated 70-90% stenosis, clinicians could directly recommend ICA or optimal medical therapy.
  Interventions: Diagnostic Test: Conventional Management Group
- MCG Group (Experimental): Based on MCG results, either ICA or optimal medical therapy was recommended.
  Interventions: Diagnostic Test: MCG Group

INTERVENTIONS:
Diagnostic Test: MCG Group — Based on MCG results, either ICA or optimal medical therapy was recommended.
  Arms: MCG Group
Diagnostic Test: Conventional Management Group — Treatment strategy is recommended based on stenosis severity, pre-test probability, and results of functional tests.
  Arms: Conventional Management Group

SUMMARY:
This rigorously designed randomized controlled trial aims to investigate whether Magnetocardiography (MCG) can optimize the clinical pathway, improve quality of life, and reduce healthcare costs in patients with stable coronary artery disease (SCAD) within real-world clinical settings, thereby generating evidence for the future application of MCG in clinical decision-making pathways.

Stable CAD patients with at least one major coronary vessel showing 50%-90% stenosis on coronary CTA will be enrolled based on predefined criteria. Stratified by study center and using a central web-based randomization system, participants will be allocated in a 1:1 ratio to either the **MCG-guided group** (where treatment recommendations for invasive coronary angiography [ICA] or optimal medical therapy are based on MCG results) or the **conventional management group** (where treatment strategy is based on stenosis severity, pre-test probability, and functional test results).

The study will proceed with the following evaluations:

1. Compare the proportion of patients with non-obstructive coronary artery disease on planned ICA performed within 90 days between the two groups, testing the hypothesis that this proportion is lower in the MCG-guided group.
2. Conduct telephone follow-ups at 90 days, 6 months, and 12 months post-enrollment to compare between-group differences in the rate of Major Adverse Cardiovascular Events (MACE), Seattle Angina Questionnaire (SAQ) scores, and total healthcare expenditures during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, regardless of gender.
2. Patients with stable coronary artery disease (CAD).
3. Coronary computed tomography angiography (CCTA) shows at least one major coronary vessel (diameter ≥2.5 mm) with 50-90% stenosis. Patients with 50-69% stenosis must have typical or atypical angina; for those with 70-90% stenosis, the presence of chest pain symptoms is not required.

   *Note: Chest pain is characterized by the following three features:* *(1) Chest discomfort lasting less than 15 minutes;* *(2) Precipitated by physical exertion or emotional stress;* *(3) Relieved by rest or nitrates.* *Based on these, angina is classified as:*
   * *Typical angina: all 3 features are present;*
   * *Atypical angina: 2 features are present;*
   * *Non-anginal chest pain: 1 or no feature is present.*
4. Willing to participate in the study and provide written informed consent.

Exclusion Criteria:

1. Previous myocardial infarction, PCI, CABG, or coronary angiography indicating stenosis ≥50% in a major vessel.
2. CCTA indicating left main coronary artery stenosis >50% and/or three-vessel disease.
3. History of cardiac dysfunction (≥ NYHA Class III), severe congenital heart disease, valvular heart disease, or cardiomyopathy.
4. Complex arrhythmias, such as frequent atrial premature beats, ventricular premature beats, atrial fibrillation, atrial flutter, etc.
5. History of metal implant placement (including mechanical valves, pacemakers, orthopedic internal fixation plates, drug pumps, etc.).
6. Claustrophobia.
7. Severe thoracic deformity.
8. Active bleeding.
9. Any disease with an expected survival of less than 1 year.
10. Completion of any of the following tests prior to enrollment: exercise ECG, stress echocardiography, stress SPECT, or stress CMR.
11. Any other condition where the investigator considers the patient unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with non-obstructive coronary artery disease on invasive coronary angiography (ICA) | From randomization through day 90 after enrollment.
  Compare the proportion of patients with non-obstructive coronary artery disease on planned invasive coronary angiography (ICA) performed within 90 days between the MCG-guided group and the conventional management group, where non-obstructive disease is defined as coronary stenosis <70% or an invasive fractional flow reserve (FFR) value ≥0.8.

SECONDARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) Score | From randomization through month 12 after enrollment.
  Patient quality of life will be assessed using the Seattle Angina Questionnaire (SAQ) at enrollment and at 3, 6, and 12 months thereafter. The assessment covers five domains: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception.
MACE | From randomization through month 12 after enrollment.
  The occurrence of Major Adverse Cardiovascular Events (MACE) will be recorded at 3, 6, and 12 months after enrollment. MACE is defined for this study as a composite of the following: hospitalization for unstable angina, unplanned revascularization beyond 90 days, non-fatal myocardial infarction (MI), and cardiac death.
Healthcare Expenditure | From randomization through month 12 after enrollment.
  Total healthcare expenditures will be collected via telephone follow-up at 7 days, 3 months, 6 months, and 12 months after enrollment.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Air Force Medical Center, People's Liberation Army of China, Beijing, Beijing Municipality
  - Beijing United Family Hospital, Beijing, Beijing Municipality
  - 首都医科大学附属北京安贞医院, Beijing, Beijing Municipality
  - The Third People's Hospital of Chengdu, Chengdu, Sichuan
  - Urumqi Friendship Hospital, Ürümqi, Xinjiang Uygur Autonomous Region

IPD SHARING:
Plan to Share IPD: Yes
The original database will be public one year after the end of the study by uploading the EXECL electronic database.
Supporting Information: Study Protocol, ICF
Time Frame: The raw data will be made publicly available starting 1 year after study completion and will remain accessible for a period of 5 years.
Access Criteria: Physicians in the relevant field may access the Individual Participant Data (IPD) and supporting information. The study protocol, informed consent forms, and raw data are available upon request via email.
URL: https://www.anzhen.org.cn/